CLINICAL TRIAL: NCT01234948
Title: Oral Malodour and Periodontal Disease-related Parameters. Clinical and Real-time PCR Findings
Brief Title: Oral Malodour and Periodontal Disease-related Parameters
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Dr Danae A. Apatzidou, Dental School, Aristotle University of Thessaloniki
Other Study IDs: self funded
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Halitosis; Periodontitis; Gingivitis
Keywords: Halitosis; VSC; Periodontitis; Gingivitis; Putative periodontal pathogens; Real-time PCR
MeSH Terms: conditions — Halitosis; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The tongue coating was collected with repeated strokes under relative pressure, using a sterile plastic microbiology loop of 10μl capacity from the terminal sulcus to the apex of the tongue. Samples were stored on ice in 1.5ml sterile Eppendorf tubes containing 0.4ml purified H2O. After vortex mixing for 30 seconds to evenly disperse the material the samples were stored at -70oC until required. The laboratory analysis was performed blind. Once thawed the tongue specimen was vortex mixed for 30 seconds and an aliquot was taken for subsequent use in the real-time PCR analysis. Lysates of samples were prepared by boiling the aliquot for 10 minutes after puncturing the cap with a fine sterile needle to prevent pressure build up.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chronic periodontitis patients: Chronic periodontitis patients had at least one site per quadrant with clinical probing depth (CPD) > 5mm and radiographic evidence of bone loss
- Generalised chronic gingivitis patients: Generalised chronic gingivitis patients presented with bleeding on probing (BOP) at > 30% of sites, CPDs < 4mm and no evidence of bone loss
- Periodontally healthy subjects: Healthy subjects had < 10% sites with BOP and no sites with CPD > 3mm

SUMMARY:
The primary aim of the current study was to determine the association between halitosis detection (presence or absence) and periodontal status in non-smoking subjects, and also assess whether halitosis recordings were related to periodontal clinical parameters, tongue coating and quantities of two putative periodontal pathogens on the posterior region of the tongue determined by real-time PCR. Secondary, halitosis recordings were compared among subjects with chronic periodontitis, chronic generalized gingivitis and periodontal health.

DETAILED DESCRIPTION:
A debate in the literature exists as to whether periodontitis is linked with oral malodour and this study attempts to understand the way in which periodontal disease is associated with oral malodour-related parameters.

Clinical protocol:

Seventy-eight systemically healthy non-smokers were screened for oral halitosis in the Department of Periodontology, Aristotle University of Thessaloniki, Greece. These were non-halitosis complaining subjects. After initial screening for suitability and obtaining a signed informed consent approved by the Ethics Committee of the Dental School, Aristotle University of Thessaloniki, a full-mouth periodontal charting was recorded including plaque index (PI), clinical probing depth (CPD), clinical attachment levels (CAL) and bleeding on probing (BOP) at six sites per tooth using a manual periodontal probe (Hu-Friedy XP-23/QW). The subjects that fulfilled the clinical inclusion criteria were classified as chronic periodontitis (N=28), chronic generalised gingivitis (N=23) or healthy individuals (27) and were further clinically and microbiologically monitored.

Assessment of tongue coating:

The Winkel Tongue Coating Index (Winkel et al., 2003) was visually determined by dividing the dorsum of the tongue into sextants. A score between zero and two was given to each sextant according to the amount of deposits and these scores were added giving a total ranging from zero to 12.

Collection of tongue sample:

A specimen was collected from the rear of the tongue dorsum for quantitative analysis of two putative periodontal pathogens, Porphyromonas gingivalis and Fusobacterium nucleatum, by real-time PCR.

In order to avoid interference of bleeding on probing and tongue sampling with the organoleptic assessments and primarily with the evaluation of the tongue odour, subjects were recalled on a second visit at the same time of the day and within a period of four days for oral malodour assessment. Within this short time interval, participants were asked not to change their routine dietary and oral hygiene habits except for 48 hours prior to the next visit when the halitosis assessments were carried out (Roldán et al., 2003; Donaldson et al., 2007). Written instructions were given to each participant regarding food and drink consumption and oral hygiene habits. In more detail, spicy food, onion, garlic, alcohol and mouthwashes were avoided 48 prior to the examination. On the morning of evaluation coffee, mints, chewing gum, oral hygiene practices, scented cosmetics or aftershave lotion were avoided. Consumption of water and oral rinses with water were allowed at least two hours prior to the odour assessment. In a similar manner, the judge who carried out the organoleptic assessments of oral malodour followed the same instructions as the participants for 24 hours before undertaking the examinations.

Oral malodour assessment:

* The Halimeter® (Halimeter® RH-17, Interscan Corporation, Chatsworth, CA, USA) was used to measure the concentration of volatile sulphide compounds (VSC) in parts per billion (p.p.b.) (Rosenberg et al., 1991). The assessments were always carried out between 10.00-12.00 at the same dental chair in the clinic to minimise daily variability in the room's temperature and humidity (Liu et al., 2006);
* Organoleptic assessments (ORG) ranging from zero to five (Rosenberg et al., 1991) assessed the odour of the following parameters:

Whole mouth air (ORG1) - subjects were asked to exhale gently into a 20cm long tube through a screen, to avoid eye contact with the odour judge, who evaluated breath odour at the other end of the tube (Murata et al., 2002); Anterior region of the dorsum of tongue (ORG2) - subjects were asked to lick their wrists and wait a couple of seconds to allow the area to dry out before the odour was assessed; Posterior region of tongue (ORG3) - material was harvested from the rear of the lingual dorsum in a standardized manner using a plastic spoon; Nose air - subjects were asked to exhale through one nostril after capping the opposite nostril with their finger in order to exclude extra-oral causes that may be related to bad breath.

A calibrated single "examiner" recorded the periodontal measurements and Halimeter® readings, whereas one calibrated "judge" carried out the organoleptic assessments of halitosis. All participants were assessed by the same examiner and judge. To assure unbiased data collection the odour judge was blinded regarding the Halimeter® measurements and the clinical status of the individual. Prior to and during this investigation the odour judge and an additional odour "evaluator" were repeatedly standardized against a wide range of n-butanol solutions with intensities from 25 to 6075 parts per million (Nachnani et al., 2005; Saad et al., 2005) and also on the mouth odour of patients attending the periodontal clinic. In order to assess the reliability of the judge's ratings, the judge and the evaluator examined the mouth odour of a number of study participants without being aware of one another's score. A statistically significant correlation was found between the scores (Spearman's rho=0.64 for the odour of whole mouth air, p<0.001) (S.A.C.M.O.T., 2002). It should be noted that only the judge's assessments were used in data analysis.

Subjects were designated as halitosis positive (+) when either the organoleptic score of the whole mouth air was two or more, and/or the readings of the Halimeter® exceeded 140 p.p.b.

Real-time polymerase chain reaction:

The DNA of P. gingivalis strain W50 and F. nucleatum strain ATCC 10953 was prepared at the Dental School, University of Glasgow following the standard protocol. Briefly, P. gingivalis and F. nucleatum were grown on fastidious anaerobe agar and harvested after three to seven days. The organisms from a single agar plate were harvested with swabs and dispersed into PBS containing 0.1mM disodium EDTA (PBSE). After one washing in PBS, they were resuspended in 1ml sterile deionised water and aliquoted into two 1.5ml screw top microcaps. DNA was extracted from the organisms by placing the tubes in a boiling water bath for ten minutes. The lysate was mixed with an equal volume of phenol: chloroform: isoamyl alcohol (25:24:1; v/v/v) for five minutes. After centrifugation (13000rpm, 10min) the aqueous upper phase from each preparation was transferred to a fresh tube and mixed with one volume of chloroform: isoamyl alcohol (24:1) for five minutes. After centrifugation (13000rpm, 10min) the aqueous upper phase from each preparation was transferred to a fresh tube and 0.1 volume of 4.5M sodium acetate solution (pH 5.4) and two volumes of ethanol were added. DNA was precipitated overnight at -20oC. The DNA was pelleted by centrifugation (13000rpm, 10min) washed sequentially in 1mL of 70% ethanol, 95% ethanol and allowed to almost dry. The DNA was then dissolved in 100µl water. The nucleic acid concentration and purity was measured at a wavelength of 260 nanometres and the ratio of the absorbance at 260 and 280 nanometres was measured using a sterile quartz cuvette in a spectrophotometer.

A real-time PCR assay using the TaqMan system (Yoshida et al., 2003) was used in the current study for the quantitative analysis of the 16S rRNA of F. nucleatum and P. gingivalis in tongue coatings. Lysates of samples were prepared by boiling the aliquot for 10 minutes after puncturing the cap with a fine sterile needle to prevent pressure build up. PCR was performed at a total volume of 20μl using the Light CyclerTM Fast Start DNA Master Hybridization Probes kit (Roche Diagnostics, Manheim, Germany), 500nM each of sense and antisense primers, 200nM probe and 5μl of lysed cells. The species-specific primers and TaqMan probes used are shown in Table 1. The specificity of the amplified products and therefore of the primers was confirmed previously (Kato et al., 2005; Yoshida et al., 2003). Amplification and detection were performed with the LightCycler Sequence Detection System (Roche Diagnostics, Manheim, Germany) with the following cycle conditions, identical for both assays: 95C for 10min, and then 45 cycles of 95C for 10sec, 58C for 25sec and a final elongation at 40C for 30sec. A standard curve was plotted for each assay by using serial dilutions of known quantities of purified genomic DNA of each test organism.

Statistical methods:

The statistical null hypothesis that there is no association between halitosis detection (presence or absence) and periodontal status in non-smoking subjects was tested by logistic regression. Since the size of each clinical group was above 20 and the minimum number of halitosis positive subjects per clinical group exceeded ten, with the exception of the healthy group (nine halitosis positive subjects), the sample size was deemed adequate for the application of this statistical model (Peduzzi et al. 1996).

The association between halitosis presence or absence and clinical indices (PI, CPD, CAL, BOP, sites > 5mm CPD, WTCI) was examined using logistic regression. Spearman's rho correlation coefficient estimated the association between scale variables and also the agreement between the scores of the two odour assessors. The assumption of normality for scale variables was tested by the Shapiro Wilk test. Between groups comparisons were performed using the Kruskal-Wallis test, while pair-wise comparisons were conducted by the Mann-Whitney test with Bonferroni's adjustment of type I error.

The analysis of data was performed using the SPSS version 16.0 software and the level of statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

The clinical inclusion criteria were as follows:

(I) Chronic periodontitis patients had at least one site per quadrant with clinical probing depth (CPD) > 5mm and radiographic evidence of bone loss; (II) Generalised chronic gingivitis patients presented with bleeding on probing (BOP) at > 30% of sites, CPDs < 4mm and no evidence of bone loss; (III) Healthy subjects had < 10% sites with BOP and no sites with CPD > 3mm.

Exclusion Criteria:

Less than 20 teeth, smoking (during the previous year), presence of any systemic disease (e.g. diabetes mellitus, gastrointestinal disorders, etc.) including ENT complications, prescribed medication that can cause xerostomia based on the Greek National Formulary of drugs, full and/or partial dentures, heavily restored dentition, large carious cavities that can trap food remnants, pathology of the oral tissues (pericoronitis, dental / periodontal abscess, etc), antibiotic therapy within three months of recruitment, periodontal treatment within the last year, pregnancy or lactation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Systemically healthy non-smokers were screened for oral halitosis in the Department of Periodontology, Aristotle University of Thessaloniki, Greece.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Halitosis presence | At a single time point
  Subjects were designated as halitosis positive (+) when either the organoleptic score of the whole mouth air was two or more, and/or the readings of the Halimeter® exceeded 140 p.p.b.

SECONDARY OUTCOMES:
Tongue coating | At a single time point
  Assessment of tongue coating:
  The Winkel Tongue Coating Index (Winkel et al., 2003) was visually determined by dividing the dorsum of the tongue into sextants. A score between zero and two was given to each sextant according to the amount of deposits and these scores were added giving a total ranging from zero to 12.
Putative periodontal pathogens | At a single time point
  A specimen was collected from the rear of the tongue dorsum for quantitative analysis of two putative periodontal pathogens, P. gingivalis and F. nucleatum, by real-time PCR.
Periodontal clinical indices | At a single time point
  plaque index, clinical probing depth, clinical attachment levels and bleeding on probing.

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Konstantinidis, Professor, Study Chair — Department of Preventive Dentistry, Periodontology and Biology of Implants, Dental School, Aristotle University of Thessaloniki, Greece
Locations (1):
- Dental School, Aristotle University, Thessaloniki, Greece

REFERENCES:
- [Background] Donaldson AC, Riggio MP, Rolph HJ, Bagg J, Hodge PJ. Clinical examination of subjects with halitosis. Oral Dis. 2007 Jan;13(1):63-70. doi: 10.1111/j.1601-0825.2006.01248.x. PMID 17241432
- [Background] Winkel EG, Roldan S, Van Winkelhoff AJ, Herrera D, Sanz M. Clinical effects of a new mouthrinse containing chlorhexidine, cetylpyridinium chloride and zinc-lactate on oral halitosis. A dual-center, double-blind placebo-controlled study. J Clin Periodontol. 2003 Apr;30(4):300-6. doi: 10.1034/j.1600-051x.2003.00342.x. PMID 12694427
- [Background] Roldan S, Winkel EG, Herrera D, Sanz M, Van Winkelhoff AJ. The effects of a new mouthrinse containing chlorhexidine, cetylpyridinium chloride and zinc lactate on the microflora of oral halitosis patients: a dual-centre, double-blind placebo-controlled study. J Clin Periodontol. 2003 May;30(5):427-34. doi: 10.1034/j.1600-051x.2003.20004.x. PMID 12716335
- [Background] Liu XN, Shinada K, Chen XC, Zhang BX, Yaegaki K, Kawaguchi Y. Oral malodor-related parameters in the Chinese general population. J Clin Periodontol. 2006 Jan;33(1):31-6. doi: 10.1111/j.1600-051X.2005.00862.x. PMID 16367853
- [Background] Murata T, Yamaga T, Iida T, Miyazaki H, Yaegaki K. Classification and examination of halitosis. Int Dent J. 2002 Jun;52 Suppl 3:181-6. doi: 10.1002/j.1875-595x.2002.tb00921.x. PMID 12090449
- [Background] Nachnani S, Majerus G, Lenton P, Hodges J, Magallanes E. Effects of training on odor judges scoring intensity. Oral Dis. 2005;11 Suppl 1:40-4. doi: 10.1111/j.1601-0825.2005.01088.x. PMID 15752097
- [Background] Saad S, Greenman J, Duffield J, Sudlow K. Use of n-butanol as an odorant to standardize the organoleptic scale of breath odour judges. Oral Dis. 2005;11 Suppl 1:45-7. doi: 10.1111/j.1601-0825.2005.01089.x. PMID 15752098
- [Background] Aaronson N, Alonso J, Burnam A, Lohr KN, Patrick DL, Perrin E, Stein RE. Assessing health status and quality-of-life instruments: attributes and review criteria. Qual Life Res. 2002 May;11(3):193-205. doi: 10.1023/a:1015291021312. PMID 12074258
- [Background] Yoshida Y, Suzuki N, Nakano Y, Shibuya K, Ogawa Y, Koga T. Distribution of Actinobacillus actinomycetemcomitans serotypes and Porphyromonas gingivalis in Japanese adults. Oral Microbiol Immunol. 2003 Jun;18(3):135-9. doi: 10.1034/j.1399-302x.2003.00034.x. PMID 12753462
- [Background] Kato H, Yoshida A, Awano S, Ansai T, Takehara T. Quantitative detection of volatile sulfur compound- producing microorganisms in oral specimens using real-time PCR. Oral Dis. 2005;11 Suppl 1:67-71. doi: 10.1111/j.1601-0825.2005.01096.x. PMID 15752104
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Rosenberg M, Kulkarni GV, Bosy A, McCulloch CA. Reproducibility and sensitivity of oral malodor measurements with a portable sulphide monitor. J Dent Res. 1991 Nov;70(11):1436-40. doi: 10.1177/00220345910700110801. PMID 1960254